CLINICAL TRIAL: NCT05987033
Title: A First-in-human Proof-of-concept Study With NVDX3, an Osteogenic Implant of Human Allogenic Origin, in the Treatment of Distal Radius Fractures in Adults.
Brief Title: Proof-of-concept Study With NVDX3 for Treatment of Distal Radius Fractures.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novadip Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVDX3-CLN01; 2023-508321-27-00 (EU CTIS Number); 2022-002304-21 (EudraCT Number)
Record Dates: First submitted 2023-07-11; First posted 2023-08-14 (Actual); Results first posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NVDX3 implant (Experimental)
  Interventions: Drug: NVDX3

INTERVENTIONS:
Drug: NVDX3 — NVDX3 is implanted during a single surgical intervention.

SUMMARY:
Prospective, single arm, monocentric clinical study to test NVDX3 in patients suffering from distal radius fracture. NVDX3 will be implanted during a single surgical intervention.

DETAILED DESCRIPTION:
This is a prospective, single arm, monocentric first-in-human PoC study in adult patients, suffering from a distal radius fracture, treated during the surgical intervention with NVDX3, an osteogenic implant from human allogeneic origin.

As per standard of care, patients with DRF are followed up to 3 months post-intervention. In the context of this trial, patient safety and IMP efficacy will be followed up to 12 months post-implant surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients within the age range of ≥18 years to ≤80 years.
2. Patient diagnosed with DRF with confirmed:

   1. Classification AO/ATO: C2 and C3 - Intra-articular & multifragmentation.
   2. Estimated volume of the targeted bone void should not exceed 5cc.
   3. Availability of diagnostic AP and LAT X-ray or CT scan.
3. Patient can undergo the targetted surgical intervention within 7 days post-DRF diagnosis.
4. Patient fulfills criteria for undergoing a surgical intervention.
5. Patient has understood and accepted to participate in the study according to all study procedures by signing the informed consent.

Exclusion Criteria:

1. Open DRF or closed DRF with increased infection risk.
2. Injury to the median nerve.
3. Previous fracture of the target distal radius.
4. Documented disease limiting mobility and functional assessments (eg. Grip strength test).
5. Dependency on crutches or any comparable walking aids.
6. Patient is overweight, has a BMI ≥35.
7. Presence of clinically significant infection at the target implant site or systemic infection.
8. History of allergic reaction or any anticipated hypersensitivity to any of the anticipated:

   1. Osteosynthesis materials (PEEK plate and screws).
   2. Anesthetic agents.
   3. Components of the NVDX3 implant.
9. Presence of any auto-immune disease, with exception of well controlled diabetes type-1 or II, or auto-immune thyroid disorders.
10. Positive serology for human immunodeficiency virus (HIV), HBcAb and/or HBsAg.
11. Presence of an active tumor.
12. Documented metabolic bone disease or any disorder, such as but not limited to high-risk osteoporosis, that could interfere with the bone healing and bone metabolism.
13. Chronic, ongoing, or planned use of medications that might affect bone metabolism or bone quality such as bisphosphonates, steroids, methotrexate, anticoagulants, immunosuppressants or immunotherapy.
14. Excessive smoking, history of chronic alcohol or drug abuse within the 12 months prior to screening.
15. Any history of experimental therapy with another investigational drug within 60 days prior to screening.
16. Pregnant women or women of childbearing potential (WOCBP) not agreeing to use an effective method of birth control3 during the course of the study. Note: WOCBP including peri-menopausal women who have had a menstrual period within 1 year prior to surgery have to have a negative pregnancy test before entering in the study.
17. Any other psychosocial, mental and physical condition which, in the opinion of the investigator, could interfere with the trial conduct, the patient's compliance or influence interpretation of the results.
18. Patient with historically elevated radiation exposure levels that could in the opinion of the investigator have introduced unacceptable radiation risks for the patient, when being accumulated with the radiological examinations planned in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Torsten Gerich, MD, Principal Investigator — Centre Hospitalier du Luxembourg
Locations (1):
- Centre Hospitalier de Luxembourg, Luxembourg, Luxembourg

RESULTS

PARTICIPANT FLOW:
Period: Enrollment
Arm/Group | NVDX3 Implant
Started | 11
Completed | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Implantd with NVDX3
Arm/Group | NVDX3 Implant
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Luxembourg | 10
Childbearing Potential Status [Count of Participants; unit: Participants] — Population: Women
  Participants
    number analyzed (Participants) | 8
    Childbearing potential | 2
    Surgical sterilisation | 0
    Peri-menopausal (menopausal for less than 1 year) | 0
    Postmenopausal for more than 1 year | 6
Use of Tobacco [Count of Participants; unit: Participants]
  Never | 6
  Current | 2
  Former | 2
Average daily number of cigarettes during the last 12 months [Mean (Standard Deviation); unit: number of cigarettes] — Population: Current smokers
  number of cigarettes
    number analyzed (Participants) | 2
    (all) | 9.0 (11.3)
Duration of tobacco use [Mean (Standard Deviation); unit: years] — Population: Former and current smokers
  years
    number analyzed (Participants) | 4
    (all) | 20.3 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Safety: Serious Treatment-emergent Adverse Events (TEAEs) and NVDX3-related TEAEs
Description: Number of participants with serious treatment-emergent adverse events (TEAEs) and NVDX3-related TEAEs
Time Frame: Between the beginning of the implant surgery (IS) and 12 months post-IS
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Serious TEAE | 1
  NVDX3-related TEAE | 1

2. Secondary Outcome: Safety: Serious TEAEs and NVDX3-related TEAEs
Description: Number of participants with serious TEAEs and NVDX3-related TEAEs
Time Frame: Between the beginning of IS and 6 weeks post-IS
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Serious TEAE | 0
  NVDX3-related TEAE | 1

3. Secondary Outcome: Safety: Serious TEAEs and NVDX3-related TEAEs
Description: Number of participants with serious TEAEs and NVDX3-related TEAEs
Time Frame: Beyond 6 weeks post-IS till 12 months post-IS
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Serious TEAE | 1
  NVDX3-related TEAE | 0

4. Secondary Outcome: Safety: TEAEs
Description: Number of participants with TEAEs
Time Frame: Between the beginning of IS and 6 weeks post-IS Beyond 6 weeks post-IS till 12 months post-IS Between the beginning of IS and 12 months post-IS
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Between the beginning of IS and 6 weeks post-IS | 7
  Beyond 6 weeks post-IS till 12 months post-IS | 8
  Between the beginning of IS and 12 months post-IS | 10

5. Secondary Outcome: Safety: Related and Unexpected TEAEs and Serious TEAEs
Description: Number of participants with related and unexpected TEAEs and serious TEAEs
Time Frame: Between the beginning of IS and 12 months post-IS
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  NVDX3-related TEAE | 1
  NVDX3-related Serious TEAE | 0
  Unexpected TEAE | 10
  Unexpected Serious TEAE | 1

6. Secondary Outcome: Safety: TEAEs of Special Interest
Description: Number of participants with TEAEs of Special Interest
Time Frame: Between the beginning of IS and 12 months post-IS
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants | 1

7. Secondary Outcome: Efficacy: Radiological Assessments on Computed Tomography (CT) Data - Evaluation of Bone Formation
Description: Radiological assessments on Computed Tomography data (CT) using the extended Lane and Sandhu Scoring tool (eLSS) compared to HD: evaluation of bone formation
Time Frame: At 3 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
Participants
  Up to 25% of the longitudinal gap filled | 0
  Up to 50% of the longitudinal gap filled | 0
  Up to 75% of the longitudinal gap filled | 2
  Up to 100% of the longitudinal gap filled | 6
  100% of the longitudinal gap filled | 1

8. Secondary Outcome: Efficacy: Radiological Assessments on Computed Tomography (CT) Data - Evaluation of Bone Formation
Description: as for outcome 7
Time Frame: At 12 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
Participants
  Up to 25% of the longitudinal gap filled | 0
  Up to 50% of the longitudinal gap filled | 0
  Up to 75% of the longitudinal gap filled | 0
  Up to 100% of the longitudinal gap filled | 0
  Bone formation : 100% of the longitudinal gap filled | 9

9. Secondary Outcome: Efficacy: Radiological Assessments on Computed Tomography (CT) Data - Evaluation of Bone Union
Description: Radiological assessments on Computed Tomography data (CT) using the extended Lane and Sandhu Scoring tool (eLSS) compared to HD: evaluation of bone union
Time Frame: At 3 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
Participants
  Up to 25% of the transverse gap filled | 1
  Up to 50% of the transverse gap filled | 1
  Up to 75% of the transverse gap filled | 3
  Up to 100% of the transverse gap filled | 3
  100% of the transverse gap filled | 1

10. Secondary Outcome: Efficacy: Radiological Assessments on Computed Tomography (CT) Data - Evaluation of Bone Union
Description: as for outcome 9
Time Frame: At 12 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
Participants
  Up to 25% of the transverse gap filled | 0
  Up to 50% of the transverse gap filled | 0
  Up to 75% of the transverse gap filled | 0
  Up to 100% of the transverse gap filled | 1
  100% of the transverse gap filled | 8

11. Secondary Outcome: Efficacy: Radiological Assessments on Computed Tomography (CT) Data - Evaluation of Bone Remodelling
Description: Radiological assessments on Computed Tomography data (CT) using the extended Lane and Sandhu Scoring tool (eLSS) compared to HD: evaluation of bone remodelling
Time Frame: At 3 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
Participants
  No evidence of remodelling against the baseline | 1
  Possible remodelling of intramedullary canal | 6
  Full remodelling of the intramedullary canal and cortex | 2

12. Secondary Outcome: Efficacy: Radiological Assessments on Computed Tomography (CT) Data - Evaluation of Bone Remodelling
Description: Radiological assessments on Computed Tomography data (CT) using the extended Lane and Sandhu Scoring tool (eLSS) compared to HD: evaluation of bone remodelling
  The total eLSS score is the sum of three individual components: bone formation, defined as filling of the longitudinal gap, is scored from 0-5 points; bone union, defined as filling of the transverse gap, is scored from 0-5 points; and bone remodeling, defined as the appearance of continuous bone architecture (trabecula and cortex) within the new bone formed in the defect, is scored from 0-2. The eLSS therefore has a score range of 0-12 points, with higher scores indicating better bone healing.
Time Frame: At 12 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
Participants
  No evidence of remodelling against the baseline | 0
  Possible remodelling of intramedullary canal | 0
  Full remodelling of the intramedullary canal and cortex | 9

13. Secondary Outcome: Efficacy: Radiological Assessments on Computed Tomography (CT) Data - Evaluation of Total Extended Lane and Sandhu Score
Description: Radiological assessments on Computed Tomography data (CT) using the extended Lane and Sandhu Scoring tool (eLSS) compared to HD: evaluation of Total extended Lane and Sandhu Score
  The total eLSS score is the sum of three individual components: bone formation, defined as filling of the longitudinal gap, is scored from 0-5 points; bone union, defined as filling of the transverse gap, is scored from 0-5 points; and bone remodeling, defined as the appearance of continuous bone architecture (trabecula and cortex) within the new bone formed in the defect, is scored from 0-2. The eLSS therefore has a score range of 0-12 points, with higher scores indicating better bone healing.
Time Frame: At 3 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
score on a scale | 8.2 (2.2)

14. Secondary Outcome: Efficacy: Radiological Assessments on Computed Tomography (CT) Data - Evaluation of Total Extended Lane and Sandhu Score
Description: as for outcome 13
Time Frame: At 12 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
score on a scale | 11.9 (0.3)

15. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Formation
Description: Radiological assessments on X-ray using the extended Lane and Sandhu Scoring tool (eLSS) compared to HD: evaluation of bone formation
Time Frame: At 2 weeks post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Up to 25% of the longitudinal gap filled | 10
  Up to 50% of the longitudinal gap filled | 0
  Up to 75% of the longitudinal gap filled | 0
  Up to 100% of the longitudinal gap filled | 0
  100% of the longitudinal gap filled | 0

16. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Formation
Description: as for outcome 15
Time Frame: At 6 weeks post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Up to 25% of the longitudinal gap filled | 0
  Up to 50% of the longitudinal gap filled | 5
  Up to 75% of the longitudinal gap filled | 4
  Up to 100% of the longitudinal gap filled | 1
  100% of the longitudinal gap filled | 0

17. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Formation
Description: as for outcome 15
Time Frame: At 3 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Up to 25% of the longitudinal gap filled | 0
  Up to 50% of the longitudinal gap filled | 1
  Up to 75% of the longitudinal gap filled | 1
  Up to 100% of the longitudinal gap filled | 7
  100% of the longitudinal gap filled | 1

18. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Formation
Description: as for outcome 15
Time Frame: At 6 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Up to 25% of the longitudinal gap filled | 0
  Up to 50% of the longitudinal gap filled | 0
  Up to 75% of the longitudinal gap filled | 1
  Up to 100% of the longitudinal gap filled | 1
  100% of the longitudinal gap filled | 8

19. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Formation
Description: Radiological assessments on X-ray data using the extended Lane and Sandhu Scoring tool (eLSS) compared to HD: evaluation of bone formation
Time Frame: At 12 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
Participants
  Up to 25% of the longitudinal gap filled | 0
  Up to 50% of the longitudinal gap filled | 0
  Up to 75% of the longitudinal gap filled | 0
  Up to 100% of the longitudinal gap filled | 0
  Bone formation : 100% of the longitudinal gap filled | 9

20. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Union
Description: Radiological assessments on X-ray using the extended Lane and Sandhu Scoring tool (eLSS) compared to HD: evaluation of bone union
Time Frame: At 2 weeks post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Up to 25% of the transverse gap filled | 10
  Up to 50% of the transverse gap filled | 0
  Up to 75% of the transverse gap filled | 0
  Up to 100% of the transverse gap filled | 0
  100% of the transverse gap filled | 0

21. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Union
Description: as for outcome 20
Time Frame: At 6 weeks post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Up to 25% of the transverse gap filled | 2
  Up to 50% of the transverse gap filled | 6
  Up to 75% of the transverse gap filled | 2
  Up to 100% of the transverse gap filled | 0
  100% of the transverse gap filled | 0

22. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Union
Description: as for outcome 20
Time Frame: At 3 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Up to 25% of the transverse gap filled | 1
  Up to 50% of the transverse gap filled | 0
  Up to 75% of the transverse gap filled | 5
  Up to 100% of the transverse gap filled | 3
  100% of the transverse gap filled | 1

23. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Union
Description: as for outcome 20
Time Frame: At 6 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  Up to 25% of the transverse gap filled | 1
  Up to 50% of the transverse gap filled | 0
  Up to 75% of the transverse gap filled | 0
  Up to 100% of the transverse gap filled | 5
  100% of the transverse gap filled | 4

24. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Union
Description: as for outcome 20
Time Frame: At 12 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
Participants
  Up to 25% of the transverse gap filled | 0
  Up to 50% of the transverse gap filled | 0
  Up to 75% of the transverse gap filled | 0
  Up to 100% of the transverse gap filled | 1
  100% of the transverse gap filled | 8

25. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Remodelling
Description: Radiological assessments on X-ray using the extended Lane and Sandhu Scoring tool (eLSS) compared to HD: evaluation of bone remodelling
Time Frame: At 2 weeks post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  No evidence of remodelling against the baseline | 10
  Possible remodelling of intramedullary canal | 0
  Full remodelling of the intramedullary canal and cortex | 0

26. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Remodelling
Description: as for outcome 25
Time Frame: At 6 weeks post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  No evidence of remodelling against the baseline | 2
  Possible remodelling of intramedullary canal | 8
  Full remodelling of the intramedullary canal and cortex | 0

27. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Remodelling
Description: as for outcome 25
Time Frame: At 3 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  No evidence of remodelling against the baseline | 1
  Possible remodelling of intramedullary canal | 7
  Full remodelling of the intramedullary canal and cortex | 2

28. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Remodelling
Description: as for outcome 25
Time Frame: At 6 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
Participants
  No evidence of remodelling against the baseline | 1
  Possible remodelling of intramedullary canal | 0
  Full remodelling of the intramedullary canal and cortex | 9

29. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Bone Remodelling
Description: as for outcome 25
Time Frame: At 12 months post-IS
Population: Number of patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
Participants
  No evidence of remodelling against the baseline | 0
  Possible remodelling of intramedullary canal | 0
  Full remodelling of the intramedullary canal and cortex | 9

30. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Total Extended Lane and Sandhu Score
Description: Radiological assessments on X-ray using the extended Lane and Sandhu Scoring tool (eLSS) compared to HD: evaluation of Total extended Lane and Sandhu Score
  The eLSS was also applied for assessment of X-ray images to support findings from CT images reflecting radiological healing over the 12-month study period. As described above, the total eLSS score is the sum of three individual components: bone formation (0-5 points), bone union (0-5 points), and bone remodeling, (0-2 points). The eLSS therefore has a score range of 0-12 points with higher scores indicating better bone healing.
Time Frame: At 2 weeks post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale | 2.0 (0.0)

31. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Total Extended Lane and Sandhu Score
Description: as for outcome 30
Time Frame: At 6 weeks post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale | 5.4 (1.5)

32. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Total Extended Lane and Sandhu Score
Description: as for outcome 30
Time Frame: At 3 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale | 8.2 (2.3)

33. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Total Extended Lane and Sandhu Score
Description: as for outcome 30
Time Frame: At 6 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale | 10.6 (2.4)

34. Secondary Outcome: Efficacy: Radiological Assessments on X-ray Data - Evaluation of Total Extended Lane and Sandhu Score
Description: as for outcome 30
Time Frame: At 12 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
score on a scale | 11.9 (0.3)

35. Secondary Outcome: Efficacy: Clinical Assessments - Grip Strength
Description: Grip strength measure with a hydraulic hand dynamometer, difference from normal (Fraction of the Strength on the Uninjured Side)
Time Frame: At 2 weeks post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
percentage
  Actual values | 26.1 (13.8)
  Change from baseline: number analyzed (Participants) | 9
  Change from baseline | 25.0 (14.6)

36. Secondary Outcome: Efficacy: Clinical Assessments - Grip Strength
Description: as for outcome 35
Time Frame: At 6 weeks post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
percentage
  Actual values | 38.8 (18.7)
  Change from baseline: number analyzed (Participants) | 9
  Change from baseline | 38.7 (19.9)

37. Secondary Outcome: Efficacy: Clinical Assessments - Grip Strength
Description: as for outcome 35
Time Frame: At 3 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
percentage
  Actual values | 67.4 (25.3)
  Change from baseline: number analyzed (Participants) | 9
  Change from baseline | 67.1 (27.2)

38. Secondary Outcome: Efficacy: Clinical Assessments - Grip Strength
Description: as for outcome 35
Time Frame: At 6 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
percentage
  Actual values | 81.9 (20.0)
  Change from baseline: number analyzed (Participants) | 9
  Change from baseline | 82.0 (21.0)

39. Secondary Outcome: Efficacy: Clinical Assessments - Grip Strength
Description: as for outcome 35
Time Frame: At 12 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
percentage
  Actual values | 93.3 (27.4)
  Change from baseline: number analyzed (Participants) | 8
  Change from baseline | 93.3 (29.8)

40. Secondary Outcome: Efficacy: Clinical Assessments - Modified Mayo Wrist Score (MMWS)
Description: Physician Reported Modified Mayo Wrist Score, total score The physician-reported MMWS is a clinical assessment that evaluates dimensions of pain, patient satisfaction, range of motion, and grip strength each on a scale of 0-25 points. The total score ranges from 0-100 points with higher scores indicating a better result.
Time Frame: At Hospital Discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
score on a scale | 36.7 (8.3)

41. Secondary Outcome: Efficacy: Clinical Assessments - Modified Mayo Wrist Score (MMWS)
Description: as for outcome 40
Time Frame: At 2 weeks post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale | 45.0 (14.7)

42. Secondary Outcome: Efficacy: Clinical Assessments - Modified Mayo Wrist Score (MMWS)
Description: as for outcome 40
Time Frame: At 6 weeks post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale | 44.5 (15.9)

43. Secondary Outcome: Efficacy: Clinical Assessments - Modified Mayo Wrist Score (MMWS)
Description: as for outcome 40
Time Frame: At 3 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale | 69.0 (17.9)

44. Secondary Outcome: Efficacy: Clinical Assessments - Modified Mayo Wrist Score (MMWS)
Description: as for outcome 40
Time Frame: At 6 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale | 76.5 (22.0)

45. Secondary Outcome: Efficacy: Clinical Assessments - Modified Mayo Wrist Score (MMWS)
Description: as for outcome 40
Time Frame: At 12 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
score on a scale | 81.1 (22.2)

46. Secondary Outcome: Efficacy: Clinical Assessments - Patient-rated Wrist Evaluation (PRWE)
Description: PRWE total score
  The PRWE consists of two subscales: the pain subscale, which contains 5 items each rated from 0 (no pain) to 10 (worst pain ever) for a total of 50 points, and the function subscale, which contains 10 items divided into specific activities (6 items) and usual activities (4 items), each rated on a scale from 0 (no difficulty) to 10 (so difficult it cannot be done). The function score is divided by 2 and added to the pain score for a total score ranges of 0-100, with lower scores indicating less wrist pain and disability.
Time Frame: At 2 weeks post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale
  Actual value | 58.4 (19.92)
  Change from baseline: number analyzed (Participants) | 9
  Change from baseline | -19.83 (21.35)

47. Secondary Outcome: Efficacy: Clinical Assessments - Patient-rated Wrist Evaluation (PRWE)
Description: as for outcome 46
Time Frame: At 6 weeks post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
score on a scale
  Actual value | 30.89 (22.33)
  Change from baseline: number analyzed (Participants) | 8
  Change from baseline | -47.88 (22.26)

48. Secondary Outcome: Efficacy: Clinical Assessments - Patient-rated Wrist Evaluation (PRWE)
Description: as for outcome 46
Time Frame: At 3 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale
  Actual value | 26.85 (23.51)
  Change from baseline: number analyzed (Participants) | 9
  Change from baseline | -48.63 (22.14)

49. Secondary Outcome: Efficacy: Clinical Assessments - Patient-rated Wrist Evaluation (PRWE)
Description: as for outcome 46
Time Frame: At 6 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale
  Actual value | 19.10 (24.99)
  Change from baseline: number analyzed (Participants) | 9
  Change from baseline | -57.39 (26.19)

50. Secondary Outcome: Efficacy: Clinical Assessments - Patient-rated Wrist Evaluation (PRWE)
Description: as for outcome 46
Time Frame: At 12 months post-IS
Population: Number of patients with assessments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
score on a scale
  Actual value | 13.44 (19.13)
  Change from baseline: number analyzed (Participants) | 8
  Change from baseline | -63.31 (19.06)

51. Secondary Outcome: Efficacy: NRS-pain
Description: NRS-pain score. NRS-pain is a patient-reported instrument for evaluating pain in clinical studies. Pain at time of the patient's visit at site was assessed on a numerical scale from 0 (no pain) to 10 (worst pain imaginable).
Time Frame: At hospital discharge
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale
  Actual value | 3.0 (1.6)
  Change from baseline | -1.5 (3.1)

52. Secondary Outcome: Efficacy: NRS-pain
Description: as for outcome 51
Time Frame: At 2 weeks post-IS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale
  Actual value | 1.9 (1.7)
  Change from baseline | -2.6 (3.1)

53. Secondary Outcome: Efficacy: NRS-pain
Description: as for outcome 51
Time Frame: At 6 weeks post-IS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale
  Actual value | 1.7 (1.8)
  Change from baseline | -2.8 (3.2)

54. Secondary Outcome: Efficacy: NRS-pain
Description: as for outcome 51
Time Frame: At 3 months post-IS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale
  Actual value | 1.6 (2.0)
  Change from baseline | -2.9 (3.7)

55. Secondary Outcome: Efficacy: NRS-pain
Description: as for outcome 51
Time Frame: At 6 months post-IS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 10
score on a scale
  Actual value | 1.2 (2.4)
  Change from baseline | -3.3 (2.2)

56. Secondary Outcome: Efficacy: NRS-pain
Description: as for outcome 51
Time Frame: At 12 months post-IS
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | NVDX3 Implant
Number analyzed (Participants) | 9
score on a scale
  Actual value | 1.2 (2.0)
  Change from baseline | -3.1 (3.0)

ADVERSE EVENTS:
Time Frame: From from the beginning of implant surgery (IS) till 12 months post-IS
Description: Including abnormal safety laboratory results and abnormal vital signs
Arm/Group | NVDX3 Implant
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NVDX3 Implant (N=10)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NVDX3 Implant (N=10)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Peripheral swelling (General disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3)
Fracture pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Pulpitis dental (Infections and infestations) | 1 (1)
Platelet count increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Electrocardiogram abnormal (Investigations) | 2 (2)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint noise (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Itching scar (Skin and subcutaneous tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-06-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT05987033/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT05987033/SAP_001.pdf